CLINICAL TRIAL: NCT04678167
Title: Evaluation of the Efficacy of BOARDING RING Glasses in the Treatment of Vestibular Neuritis
Brief Title: Boarding Ring Glasses Versus Placebo Glasses or Not Glasses in the Treatment of Vestibular Neuritis
Acronym: NEVRING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 29BRC20.0040
Record Dates: First submitted 2020-10-02; First posted 2020-12-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Vestibular Neuritis
Keywords: vestibular hyporeflexia; rotational vertigo; horizontal-rotational nystagmus
MeSH Terms: conditions — Vestibular Neuronitis | interventions — Caloric Tests

STUDY DESIGN:
Intervention Model Description: The randomization list is established by the Brest CHRU data management unit before the start of the trial. Based on a ratio (1:1:1) with stratification on the center.
Who Masked: Investigator
Masking Description: Only the investigator carrying out the follow-up consultations is blind.
  After examination by the ENT specialist (otorhinolaryngologist) who will diagnose vestibular neuritis, the patient will be randomized into one of three groups. The clinical follow-up will be performed by another practitioner, who will not know in which arm the patient is included (the patient will come to the consultation without his glasses). Only the practitioner who realized the randomization and the patient will have information about the arm in which they are located.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Boarding ring glasses (Experimental): Realization of the following examinations WITH Boarding ring glasses :
  * caloric tests,
  * measurement of the speed of Nystagmus,
  * angle of deviation in Fukuda,
  * Alexander's degree of nystagmus,
  * EHTEV and EEV questionnaires,
  * anxiety VAS
  Interventions: Diagnostic Test: Caloric test; Diagnostic Test: Measurement of the speed of Nystagmus; Diagnostic Test: Angle of deviation at Fukuda; Diagnostic Test: Alexander's degree of nystagmus; Other: EHTEV questionnaire; Other: EEV questionnaire; Other: anxiety VAS
- Placebo glasses (Placebo Comparator): Realization of the following examinations WITH Placebo glasses :
  * caloric tests,
  * measurement of the speed of Nystagmus,
  * angle of deviation in Fukuda,
  * Alexander's degree of nystagmus,
  * EHTEV and EEV questionnaires,
  * anxiety VAS
  Interventions: Diagnostic Test: Caloric test; Diagnostic Test: Measurement of the speed of Nystagmus; Diagnostic Test: Angle of deviation at Fukuda; Diagnostic Test: Alexander's degree of nystagmus; Other: EHTEV questionnaire; Other: EEV questionnaire; Other: anxiety VAS
- No glasses (Other): Realization of the following examinations WITHOUT glasses :
  * caloric tests,
  * measurement of the speed of Nystagmus,
  * angle of deviation in Fukuda,
  * Alexander's degree of nystagmus,
  * EHTEV and EEV questionnaires,
  * anxiety VAS
  Interventions: Diagnostic Test: Caloric test; Diagnostic Test: Measurement of the speed of Nystagmus; Diagnostic Test: Angle of deviation at Fukuda; Diagnostic Test: Alexander's degree of nystagmus; Other: EHTEV questionnaire; Other: EEV questionnaire; Other: anxiety VAS

INTERVENTIONS:
Diagnostic Test: Caloric test — Lying, patientwill be placed so that he can introduce water (hot then cold) into his external ear canal. It is the reaction of the vestibular system (sensory organ responsible for balance) which is then measured with a helmet placed over his eyes and which measures the nystagmus (movement of the eye) which reflects vestibular activity.
  Other Names: Barany test
Diagnostic Test: Measurement of the speed of Nystagmus — A helmet with an infrared camera will be placed in front of patient eyes. This will allow visualizing on screen and measuring eye movements spontaneous or induced in the dark by various tests.
Diagnostic Test: Angle of deviation at Fukuda — The patient will be asked to trample on the spot (30 steps) with the indexes pointed forward. In the event of vestibular asymmetry, the patient turns at a varying angle to the right or to the left. This will then measure what is called the angle of deflection of the fukuda.
Diagnostic Test: Alexander's degree of nystagmus — there are 3 degrees:
  * Degree I: nystagmus that exists only when the eyes are turned to the right.
  * Degree II: also exists when the eyes are to the right or to the front.
  * Degree Ill: exists when the eyes are on the right, front, or left
Other: EHTEV questionnaire — Handicap Scale for Balance Disorders and Vertigo
Other: EEV questionnaire — European Vertigo Assessment Questionnaire
Other: anxiety VAS — visual analog scale of anxiety

SUMMARY:
Vestibular neuritis is a brutal and continuous dizzying syndrome of peripheral (vestibular) origin without cochlear or other associated involvement. Specifically, vestibular neuritis is inflammation of the nerve that innervates the vestibular canals (the inner ear). It is characterized by the sudden onset of intense and prolonged vertigo accompanied by postural imbalance, nausea and vomiting, without hearing impairment or other neurological symptoms. Vestibular neuritis is the second cause of peripheral vertigo after benign paroxysmal positional vertigo. It represents approximately 7% of patients consulting for vertigo. The purpose of this study is to evaluate if wearing Boarding Ring glasses can be accelerated vestibular compensation.

ELIGIBILITY:
Inclusion Criteria:

* adult patients,
* patient with vestibular neuritis defined by appearance of continuous rotating vertigo with nausea
* patient with spontaneous horizonto-rotating nystagmus beating towards the healthy ear
* patient with a postural deviation towards the affected ear;
* vestibular hyporeflexia measured at the caloric tests greater than 25%
* patient who has given free, enlighten and written consent

Exclusion Criteria:

* patient with a history of vertigo of vestibular origin or with vertigo developing for more than 4 days
* patient with associated hearing loss or tinnitus
* patient with an motor ocular abnormality of central origin
* patient refusal or inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2027-03-10 (Estimated); Study Completion 2027-03-10 (Estimated)

PRIMARY OUTCOMES:
Variation of the angle of deviation at the Fukuda test between J0 and J7 (value at J0 minus value at J7). | 7 day

SECONDARY OUTCOMES:
Speed of nystagmus | 1 year
Alexander's degree of nystagmus | 1 year
  Measure of the degree of intensity of nystagmus. There are 3 degrees :
  * Degree I: nystagmus which exists only when the eyes are turned to the right.
  * Degree II: also exists when the eyes are to the right or to the front.
  * Degree Ill: exists when the eyes are on the right, front, or left.
Duration of hospitalization (for hospitalized patients) | 1 year
Anxiety visual analog scale | 1 year
  0 = no anxiety, 10 = maximum anxiety imaginable
Handicap related to Balance Disorders and Vertigo scale (EHTEV questionnaire) | 1 year
  It helps to determine the physical, emotional and functional difficulties experienced in everyday life. EHTEV questionnaire is scored on 100 points.
  The physical score from 0 to 28 points, the emotional score from 0 to 36 points and the functional score from 0 to 36 points. ( 0 = no difficulty).
European Vertigo Evaluation Scale (EEV questionnaire) | 1 year
  Makes it possible to quantify vertigo and the associated vestibular symptoms and to monitor their evolution. EEV questionnaire is scored on 20 points (0 = no symptoms, 20 = maximum symptoms)
Vestibular deficit at caloric tests | 1 year
  measures 7of nystagmus (= fluttering of the eye) which reflects vestibular activity
Variation from J0 of the angle of deviation at the Fukuda measured at J14, M1, M3, M6, M12 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe LECLERE, Dr, Principal Investigator — University Hospital, Brest
Locations (3):
- France (3):
  - CHU de Brest, Brest
  - CH Pays de Morlaix, Morlaix
  - CH de Cornouaille Quimper, Quimper

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.